CLINICAL TRIAL: NCT03828292
Title: A Phase I Open-Label, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Clinical Activity of the Antibody Drug Conjugate GSK2857916 in Japanese Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: An Open-label, Dose Escalation Study in Japanese Participants With Relapsed/Refractory Multiple Myeloma Who Have Failed Prior Anti Myeloma Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 207504
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Antibody drug conjugate; Dose-escalation; GSK2857916; Japanese; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Bortezomib; Dexamethasone; pomalidomide

STUDY DESIGN:
Intervention Model Description: Participants will receive GSK2857916 monotherapy during Part 1 (Dose escalation) of the study on a once every 21 days schedule. During Part 2, participants will receive GSK2857916 given in combination with Bortezomib/Dexamethasone on a once every 21 days schedule (Arm A) or with Pomalidomide/Dexamethasone on a once every 28 days schedule (Arm B).
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Belantamab mafodotin Monotherapy (Experimental)
  Interventions: Drug: Belantamab mafodotin
- Part 2: Arm A: Belantamab mafodotin+Bortezomib/Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Dexamethasone
- Part 2: Arm B: Belantamab mafodotin+Pomalidomide/Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered as an intravenous infusion.
Drug: Bortezomib — Bortezomib solution for injection will be administered subcutaneously.
  Arms: Part 2: Arm A: Belantamab mafodotin+Bortezomib/Dexamethasone
Drug: Dexamethasone — Dexamethasone tablets will be administered orally.
  Arms: Part 2: Arm A: Belantamab mafodotin+Bortezomib/Dexamethasone; Part 2: Arm B: Belantamab mafodotin+Pomalidomide/Dexamethasone
Drug: Pomalidomide — Pomalidomide capsules will be administered orally.
  Arms: Part 2: Arm B: Belantamab mafodotin+Pomalidomide/Dexamethasone

SUMMARY:
Belantamab mafodotin (GSK2857916) is a first in class, antibody dependent cellular cytotoxicity (ADCC) enhanced, humanized immunoglobulin G1 (IgG1) antibody-drug conjugate (ADC) which binds specifically to B cell maturation antigen (BCMA) expressed on tumor cells of all participants with multiple myeloma. This is a Phase 1, open label, dose escalation study to investigate safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity and clinical activity of GSK2857916 when given as monotherapy (Part 1) or given as combination therapy (Part 2). Dose escalation will follow a 3+3 design.

ELIGIBILITY:
Inclusion Criteria

* Provide signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 20 years or older (at the time consent is obtained).
* ECOG performance status of 0 to 2.
* Histologically or cytologically confirmed diagnosis of multiple myeloma as defined according to IMWG 2014, criteria in a participant who fulfills all of the following: has undergone stem cell transplant, or is considered transplant ineligible, Part 1: has received at least 2 prior lines of anti-myeloma drugs containing at least 1 proteasome inhibitor and at least 1 immunomodulator, Part 2: has received at least 1 prior line of anti-myeloma drugs; has demonstrated progression on, or within 60 days of completion of the last therapy.
* Has measurable disease with at least one of the following: serum M-protein >=0.5 grams per deciliter (g/dL) (>=5 grams per liter [g/L]); Urine M-protein >=200 mg/24 hours; Serum free light chain (FLC) assay: Involved FLC level >=10 mg/dL (>=100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met: Transplant was >100 days prior to study enrolment; No active infection.
* Female participants: Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breast feeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or For Part 1 and Part 2 Arm A: Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1 percent per year), preferably with low user dependency, during the treatment period and for 4 months after the last dose of GSK2857916, and 7 months from the last dose of bortezomib (only Part 2 Arm A), and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study treatment and agree to use effective contraception during the study and for 4 months after the last dose of GSK2857916, and 7 months from the last dose of bortezomib (only Part 2 Arm A); For Part 2 Arm B: Due to pomalidomide being a thalidomide analogue with risk for embryo-fetal toxicity and prescribed under a restricted distribution program, WOCBP participants will be eligible if they commit either to abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control, beginning 4 weeks prior to initiating treatment with pomalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of pomalidomide treatment. Thereafter, WOCBP participants must use a contraceptive method that is highly effective (with a failure rate of <1 percent per year) for a further 3 months, and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. Two negative pregnancy tests must be obtained prior to initiating pomalidomide therapy. The first test should be performed within 10 to 14 days and the second test within 24 hours prior to prescribing pomalidomide therapy. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Male participants: Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following from the time of first dose of study treatment until 6 months after the last dose of GSK2857916, 4 months after the last dose of bortezomib (only Part 2 Arm A), and 4 weeks after the last dose of pomalidomide (only Part 2 Arm B) to allow for clearance of any altered sperm: Refrain from donating sperm plus either: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception/barrier as detailed: Agree to use a male condom even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1 percent per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
* All prior treatment-related toxicities (defined by National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.03, must be <=Grade 1 at the time of enrolment except for alopecia. Participants with Grade 2 peripheral neuropathy can be enrolled into Part 1 and Part 2 Arm B but not into Part 2 Arm A.
* Adequate Organ System Function. Exclusion Criteria
* Systemic anti-tumor-therapy within 14 days, or plasmapheresis within 7 days prior to the first dose of study treatment.
* Symptomatic amyloidosis, active 'polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes' (POEMS) syndrome, active plasma cell leukemia at the time of screening.
* Use of an investigational drug within 14 days or 5 half-lives, whichever is shorter, preceding the first dose of study treatment. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study treatment. Prior BCMA targeted therapy.
* History of an allogeneic stem cell transplant.
* Current use of prohibited medications/device or planned use of any of these during the study period.
* Current corneal epithelial disease except mild punctate keratopathy
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from multiple myeloma are eligible, provided they fulfil the required criteria.
* Evidence of active mucosal or internal bleeding.
* Any major surgery within the last 4 weeks.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Active infection requiring treatment (antibiotic, antiviral, or antifungal treatment).
* Evidence of severe or uncontrolled systemic diseases.
* Malignancies other than disease under study are excluded, except for any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the investigators and Medical Monitor, will not affect the evaluation of the effects of this clinical study treatment on the currently targeted malignancy (multiple myeloma).
* Evidence of cardiovascular risk including any of the following:

  1. Corrected QT interval Fridericia (QTcF) interval >=470 milliseconds (msecs) (the QT interval values must be corrected for heart rate by Fridericia's formula [QTcF])
  2. Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
  3. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 6 months of Screening.
  4. Class III or IV heart failure as defined by the New York Heart Association functional classification system
  5. Uncontrolled hypertension
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2857916 or any of the components of the study treatment.
* Pregnant or lactating female or female who are interrupting lactation.
* Known human Immunodeficiency virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb) or hepatitis B core antibody (HBcAb at Screening or within 3 months prior to first dose of study treatment).
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment. Participants with positive hepatitis C antibody due to prior resolved disease can only be enrolled, if a confirmatory negative hepatitis C RNA test is obtained. Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria.
* Previously diagnosed with interstitial lung disease or current complication of interstitial lung disease.

Additional Exclusion Criteria for Part 2 Arm A

* Intolerant to bortezomib or refractory to bortezomib.
* Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.
* Intolerance or contraindications to herpes zoster prophylaxis Additional Exclusion Criteria for Part 2 Arm B
* Prior pomalidomide use.
* Intolerance or contraindications to antithrombotic prophylaxis.
* Active or history of venous thromboembolism within 3 months prior to first dose of study treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Shibuya-Ku, Tokyo
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

REFERENCES:
- [Background] Sunami K, Iida S, Tsukada N, Fujii T, Kato H, Fukushima R, Wakabayashi S, Nakano H, Roy-Ghanta S, Kremer BE. DREAMM-11, Part 2: Japanese phase I trial of belantamab mafodotin combination therapies in relapsed/refractory multiple myeloma. Int J Hematol. 2025 Feb;121(2):174-186. doi: 10.1007/s12185-024-03889-8. Epub 2024 Dec 24. PMID 39718747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of two phases - Main Study Phase and Post Analysis Continued Treatment (PACT) Phase. In PACT phase those participants benefiting from drug continued to receive study drug until discontinuation or withdrawal from study.
Groups:
- Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg): Participants with Relapsed or Refractory Multiple Myeloma (RRMM) received belantamab mafodotin as 2.5 milligram (mg)/kilogram (kg) dose via intravenous (IV) infusion on Day 1 of every 21-day cycle (Q3W) maximum up to disease progression.
- Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg: Participants with RRMM received belantamab mafodotin as dose of 3.4 mg/kg via IV infusion on Day 1 of every 21-day cycle (Q3W) maximum up to disease progression.
- Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex); PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex): Participants with RRMM received belantamab mafodotin as dose of 2.5mg/kg via IV infusion on Day 1 of every 21-day cycle (Q3W) maximum up to disease progression. Bortezomib was administered subcutaneously (SC) as 1.3 mg/meter^2 (m^2) on Day 1, Day 4, Day 8, and Day 11 of every 21-day cycle maximum up to 8 cycles. Dexamethasone was administered orally as dose of 20 mg on Day 1, Day 2, Day 4, Day 5, Day 8, Day 9, Day 11, and Day 12 of every 21-day cycle maximum up to 8 cycles.
- Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex); PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex): Participants with RRMM received belantamab mafodotin at a dose of 2.5 mg/kg via IV infusion on Day 1 of each 28-day cycle in cycle 1, and at a dose of 1.9 mg/kg from cycle 2 onwards maximum up to disease progression. Along with belantamab mafodotin, Pomalidomide was administered orally as dose of 4 mg per day on Day 1 to Day 21 of 28-day cycles maximum up to disease progression. Dexamethasone orally as dose of 40 mg per day on Day 1, Day 8, Day 15, and Day 22 of each 28-day maximum up to disease progression.
Period: Main Study: Part 1 (Up to 141 Weeks)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex)
Started | 4 | 4 | 0 | 0 | 0 | 0
Completed | 4 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Period: Main Study: Part 2 (Up to 212 Weeks)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex)
Started | 0 | 0 | 3 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Transitioned to PACT | 0 | 0 | 2 | 2 | 0 | 0
Period: PACT Phase (From 212 to 286 Weeks)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex)
Started | 0 | 0 | 0 | 0 | 2 (Participant transitioned from main study phase to PACT Phase) | 2 (Participant transitioned from main study phase to PACT Phase)
Completed | 0 | 0 | 0 | 0 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) | Total
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 15
Age, Customized [Count of Participants; unit: Participants]
  20 to 76 years | 4 | 4 | 3 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 5
  Male | 3 | 2 | 2 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian- Japanese Heritage | 4 | 4 | 3 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is an Adverse Event (AE) that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 21-day DLT period and meets at least one of the DLT criteria: Grade 3 or greater febrile neutropenia lasting >48 hours (h) despite adequate treatment, Grade 4 thrombocytopenia <25,000/mm^3accompanied by clinically significant bleeding, any Grade 3 or greater non-hematologic toxicity, any Grade 3 or greater non-hematologic laboratory value if: laboratory abnormality persists for >48 h despite supportive treatment for abnormality leads to hospitalization, Grade 4 Corneal toxicity, and liver toxicity meeting pre-specified GlaxoSmithKline liver stopping criteria. DLTs were assessed by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.03.
Time Frame: Up to Day 21
Population: DLT Evaluable population included participants fulfilling the 'All Treated' population (all eligible participants who received at least 1 dose of study treatment) criteria, and those who received a complete infusion in 21- day Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Primary Outcome: Part 2: Arm A: Number of Participants With DLTs
Description: DLT is an AE that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 21-day DLT period and meets at least one of the DLT criteria: Grade 3 or greater febrile neutropenia lasting >48 hours (h) despite adequate treatment, Grade 4 thrombocytopenia <25,000/mm^3 accompanied by clinically significant bleeding, any Grade 3 or greater non-hematologic toxicity, any Grade 3 or greater non-hematologic laboratory value if: laboratory abnormality persists for >48 h despite supportive treatment or abnormality leads to hospitalization, Grade 4 Corneal toxicity, and liver toxicity meeting pre-specified GlaxoSmithKline liver stopping criteria. DLTs were assessed by NCI-CTCAE, version 4.03.
Time Frame: Up to Day 21
Population: DLT Evaluable population included participants fulfilling the 'All Treated' population criteria, and those who received a complete infusion of Belantamab Mafodotin and at least 75% of planned doses of bortezomib/dexamethasone in 21-day Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Part 2: Arm B: Number of Participants With DLTs
Description: as for outcome 2
Time Frame: Up to Day 28
Population: DLT Evaluable population included participants fulfilling the 'All Treated' population criteria, and those who received a complete infusion of Belantamab Mafodotin and at least 75% of planned doses of pomalidomide/dexamethasone in 28-day Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 4
Participants | 1

4. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; was a congenital anomaly/birth defect. SAEs are subset of AEs.
Time Frame: Up to approximately 141 weeks
Population: All Treated Population included all eligible participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  AEs | 4 | 4
  SAEs | 2 | 0

5. Primary Outcome: Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent disability/incapacity or Is a congenital anomaly/birth defect other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs.
Time Frame: Up to approximately 212 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  AEs | 3 | 4
  SAEs | 0 | 1

6. Primary Outcome: Part 1: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for clinical chemistry parameters analysis: Creatine Kinase (CK), Creatinine, Gamma Glutamyl Transferase (GGT), Magnesium, Phosphate, Potassium, Sodium, Calcium, Glucose, Urate, Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Bilirubin were graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v) 4.03. Grade (G)1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Any worst-case post baseline increases in grade along with any increase to a maximum G3 and a maximum G4 are presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population. Only those participants with data available at specified category have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Hyperglycemia, Any Grade Increase | 4 | 4
  Hyperglycemia, Increase to Grade 3 | 0 | 0
  Hyperglycemia, Increase to Grade 4 | 0 | 0
  CK, Any Grade Increase | 1 | 0
  CK, Increase to Grade 3 | 0 | 0
  CK, Increase to Grade 4 | 0 | 0
  Creatinine, Any Grade Increase | 0 | 0
  Creatinine, Increase to Grade 3 | 0 | 0
  Creatinine, Increase to Grade 4 | 0 | 0
  GGT, Any Grade Increase | 2 | 2
  GGT, Increase to Grade 3 | 1 | 2
  GGT, Increase to Grade 4 | 0 | 0
  Hypermagnesemia, Any Grade Increase | 1 | 0
  Hypermagnesemia, Increase to Grade 4 | 0 | 0
  Hypermagnesemia, Increase to Grade 3 | 0 | 0
  Hypomagnesemia, Any Grade Increase | 1 | 1
  Hypomagnesemia, Increase to Grade 3 | 0 | 0
  Hypomagnesemia, Increase to Grade 4 | 0 | 0
  Phosphate, Any Grade Increase | 1 | 2
  Phosphate, Increase to Grade 3 | 0 | 1
  Phosphate, Increase to Grade 4 | 0 | 0
  Hyperkalemia, Any Grade Increase | 0 | 2
  Hyperkalemia, Increase to Grade 3 | 0 | 1
  Hyperkalemia, Increase to Grade 4 | 0 | 0
  Hypokalemia, Any Grade Increase | 2 | 2
  Hypokalemia, Increase to Grade 3 | 0 | 1
  Hypokalemia, Increase to Grade 4 | 0 | 0
  Hypernatremia, Any Grade Increase | 1 | 0
  Hypernatremia, Increase to Grade 3 | 0 | 0
  Hypernatremia, Increase to Grade 4 | 0 | 0
  Hypoglycemia, Any Grade Increase | 2 | 1
  Hypoglycemia, Increase to Grade 3 | 0 | 0
  Hypoglycemia, Increase to Grade 4 | 0 | 0
  Hyponatremia, Any Grade Increase | 1 | 3
  Hyponatremia, Increase to Grade 3 | 0 | 1
  Hyponatremia, Increase to Grade 4 | 0 | 0
  Hyperuricemia, Any Grade Increase | 0 | 0
  Hyperuricemia, Increase to Grade 3 | 0 | 0
  Hyperuricemia, Increase to Grade 4 | 0 | 0
  ALT, Any Grade Increase | 3 | 3
  ALT, Increase to Grade 3 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0
  Albumin, Any Grade Increase | 2 | 1
  Albumin, Increase to Grade 3 | 0 | 0
  Albumin, Increase to Grade 4 | 0 | 0
  ALP, Any Grade Increase | 2 | 1
  ALP, Increase to Grade 3 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0
  AST, Any Grade Increase | 4 | 4
  AST, Increase to Grade 3 | 1 | 1
  AST, Increase to Grade 4 | 0 | 0
  Bilirubin, Any Grade Increase | 1 | 1
  Bilirubin, Increase to Grade 3 | 0 | 0
  Bilirubin, Increase to Grade 4 | 0 | 0
  Hypercalcemia, Any Grade Increase | 1 | 1
  Hypercalcemia, Increase to Grade 3 | 0 | 0
  Hypercalcemia, Increase to Grade 4 | 0 | 0
  Hypocalcemia, Any Grade Increase | 2 | 0
  Hypocalcemia, Increase to Grade 3 | 0 | 0
  Hypocalcemia, Increase to Grade 4 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of clinical chemistry parameters: C Reactive Protein, Chloride, Direct Bilirubin (DB), Lactate Dehydrogenase, Protein and Urea. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE v4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population. Participants are counted twice if the participant has values that changed "Decreased to Low" and "Increased to High", so the sum of the percentages may not add to 100% for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  C Reactive Protein, Decrease to Low: number analyzed (Participants) | 4 | 3
  C Reactive Protein, Decrease to Low | 0 | 0
  C Reactive Protein, Change to Normal or No Change: number analyzed (Participants) | 4 | 3
  C Reactive Protein, Change to Normal or No Change | 2 | 1
  C Reactive Protein, Increase to High: number analyzed (Participants) | 4 | 3
  C Reactive Protein, Increase to High | 2 | 2
  Chloride, Decrease to Low | 2 | 2
  Chloride, Change to Normal or No Change | 0 | 2
  Chloride, Increase to High | 2 | 1
  Direct Bilirubin, Decrease to Low | 0 | 0
  Direct Bilirubin, Change to Normal or No Change | 4 | 3
  Direct Bilirubin, Increase to High | 0 | 1
  Lactate Dehydrogenase, Decrease to Low | 0 | 0
  Lactate Dehydrogenase, Change to Normal or No Change | 2 | 2
  Lactate Dehydrogenase, Increase to High | 2 | 2
  Protein, Decrease to Low | 1 | 2
  Protein, Change to Normal or No Change | 2 | 2
  Protein, Increase to High | 1 | 0
  Urea, Decrease to Low | 2 | 1
  Urea, Change to Normal or No Change | 1 | 2
  Urea, Increase to High | 1 | 1

8. Primary Outcome: Part 2: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for clinical chemistry parameters analysis: Creatine Kinase (CK), Creatinine, Gamma Glutamyl Transferase (GGT), Magnesium, Phosphate, Potassium, Sodium, Calcium, Glucose, Urate, Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Bilirubin were graded according to NCI-CTCAE v 4.03. G1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Any worst-case post baseline increases in grade along with any increase to a maximum G3 and a maximum G4 are presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified category have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Hyperglycemia, Any Grade Increase | 1 | 4
  Hyperglycemia, Increase to Grade 3 | 0 | 0
  Hyperglycemia, Increase to Grade 4 | 0 | 0
  Hypoglycemia, Any Grade Increase | 1 | 1
  Hypoglycemia, Increase to Grade 3 | 0 | 0
  Hypoglycemia, Increase to Grade 4 | 0 | 0
  ALT, Any Grade Increase | 2 | 3
  ALT, Increase to Grade 3 | 0 | 1
  ALT, Increase to Grade 4 | 0 | 0
  Albumin, Any Grade Increase | 1 | 3
  Albumin, Increase to Grade 3 | 0 | 0
  Albumin, Increase to Grade 4 | 0 | 0
  ALP, Any Grade Increase | 2 | 4
  ALP, Increase to Grade 3 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0
  AST, Any Grade Increase | 3 | 2
  AST, Increase to Grade 3 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0
  Bilirubin, Any Grade Increase | 0 | 0
  Bilirubin, Increase to Grade 3 | 0 | 0
  Bilirubin, Increase to Grade 4 | 0 | 0
  Hypercalcemia, Any Grade Increase | 0 | 0
  Hypercalcemia, Increase to Grade 3 | 0 | 0
  Hypercalcemia, Increase to Grade 4 | 0 | 0
  Hypocalcemia, Any Grade Increase | 3 | 2
  Hypocalcemia, Increase to Grade 3 | 0 | 0
  Hypocalcemia, Increase to Grade 4 | 0 | 0
  CK, Any Grade Increase: number analyzed (Participants) | 3 | 3
  CK, Any Grade Increase | 1 | 0
  CK, Increase to Grade 3: number analyzed (Participants) | 3 | 3
  CK, Increase to Grade 3 | 0 | 0
  CK, Increase to Grade 4: number analyzed (Participants) | 3 | 3
  CK, Increase to Grade 4 | 0 | 0
  Creatinine, Any Grade Increase | 1 | 1
  Creatinine, Increase to Grade 3 | 0 | 0
  Creatinine, Increase to Grade 4 | 0 | 0
  GGT, Any Grade Increase | 2 | 3
  GGT, Increase to Grade 3 | 0 | 0
  GGT, Increase to Grade 4 | 0 | 0
  Hypermagnesemia, Any Grade Increase | 0 | 0
  Hypermagnesemia, Increase to Grade 3 | 0 | 0
  Hypermagnesemia, Increase to Grade 4 | 0 | 0
  Hypomagnesemia, Any Grade Increase | 1 | 2
  Hypomagnesemia, Increase to Grade 3 | 0 | 0
  Hypomagnesemia, Increase to Grade 4 | 0 | 0
  Phosphate, Any Grade Increase | 2 | 2
  Phosphate, Increase to Grade 3 | 0 | 1
  Phosphate, Increase to Grade 4 | 0 | 0
  Hyperkalemia, Any Grade Increase | 0 | 0
  Hyperkalemia, Increase to Grade 3 | 0 | 0
  Hyperkalemia, Increase to Grade 4 | 0 | 0
  Hypokalemia, Any Grade Increase | 3 | 1
  Hypokalemia, Increase to Grade 3 | 1 | 0
  Hypokalemia, Increase to Grade 4 | 0 | 0
  Hypernatremia, Any Grade Increase | 1 | 0
  Hypernatremia, Increase to Grade 3 | 0 | 0
  Hypernatremia, Increase to Grade 4 | 0 | 0
  Hyponatremia, Any Grade Increase | 1 | 1
  Hyponatremia, Increase to Grade 3 | 0 | 0
  Hyponatremia, Increase to Grade 4 | 0 | 0
  Hyperuricemia, Any Grade Increase | 0 | 0
  Hyperuricemia, Increase to Grade 3 | 0 | 0
  Hyperuricemia, Increase to Grade 4 | 0 | 0

9. Primary Outcome: Part 2: Number of Participants With Worst-case Change Post-baseline in Clinical Chemistry Parameters
Description: as for outcome 7
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified category have been analyzed. Participants are counted twice if the participant has values that changed "Decreased to Low" and "Increased to High", so the sum of the percentages may not add to 100% for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Direct Bilirubin, Decrease to Low | 0 | 0
  Direct Bilirubin, Change to Normal or No Change | 3 | 2
  Direct Bilirubin, Increase to High | 0 | 2
  Chloride, Decrease to Low | 2 | 1
  Chloride, Change to Normal or No Change | 0 | 2
  Chloride, Increase to High | 2 | 2
  C Reactive Protein, Decrease to Low | 0 | 0
  C Reactive Protein, Change to Normal or No Change | 2 | 1
  C Reactive Protein, Increase to High | 1 | 3
  Lactate Dehydrogenase, Decrease to Low | 0 | 0
  Lactate Dehydrogenase, Change to Normal or No Change | 1 | 3
  Lactate Dehydrogenase, Increase to High | 2 | 1
  Protein, Decrease to Low | 3 | 3
  Protein, Change to Normal or No Change | 0 | 1
  Protein, Increase to High | 0 | 0
  Urea, Decrease to Low | 0 | 0
  Urea, Change to Normal or No Change | 1 | 3
  Urea, Increase to High | 2 | 1

10. Primary Outcome: Part 1: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for analysis of hematology parameters: Hemoglobin, Leukocytes, Lymphocytes, Neutrophils and Platelets were graded according to CTCAE v4.03. G1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Any worst-case post baseline increases in grade along with any increase to a maximum G3 and a maximum G4 are presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Anemia, Any Grade Increase | 1 | 2
  Anemia, Increase to Grade 3 | 0 | 1
  Anemia, Increase to Grade 4 | 0 | 0
  Hemoglobin increased, Any Grade Increase | 0 | 0
  Hemoglobin increased, Increase to Grade 3 | 0 | 0
  Hemoglobin increased, Increase to Grade 4 | 0 | 0
  Leukocytosis, Any Grade Increase | 0 | 0
  Leukocytosis, Increase to Grade 3 | 0 | 0
  Leukocytosis, Increase to Grade 4 | 0 | 0
  White blood cell decreased, Any Grade Increase | 4 | 1
  White blood cell decreased, Increase to Grade 3 | 2 | 0
  White blood cell decreased, Increase to Grade 4 | 0 | 1
  Lymphocyte count decreased, Any Grade Increase | 4 | 2
  Lymphocyte count decreased, Increase to Grade 3 | 2 | 1
  Lymphocyte count decreased, Increase to Grade 4 | 1 | 1
  Lymphocyte count increased, Any Grade Increase | 0 | 0
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0
  Neutrophils, Any Grade Increase | 4 | 3
  Neutrophils, Increase to Grade 3 | 2 | 1
  Neutrophils, Increase to Grade 4 | 0 | 0
  Platelets, Any Grade Increase | 4 | 3
  Platelets, Increase to Grade 3 | 4 | 1
  Platelets, Increase to Grade 4 | 0 | 2

11. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: Basophils, Eosinophils, Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Hemoglobin (MCH), Mean Corpuscular Volume (MCV), erythrocytes, Hematocrit, monocytes and reticulocytes. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Basophils, Decrease to Low | 0 | 0
  Basophils, Change to Normal or No Change | 4 | 4
  Basophils, Increase to High | 0 | 0
  Eosinophils, Decrease to Low | 0 | 0
  Eosinophils, Change to Normal or No Change | 3 | 4
  Eosinophils, Increase to High | 1 | 0
  MCHC, Decrease to Low | 0 | 1
  MCHC, Change to Normal or No Change | 4 | 2
  MCHC, Increase to High | 0 | 1
  MCH, Decrease to Low | 1 | 1
  MCH, Change to Normal or No Change | 3 | 3
  MCH, Increase to High | 0 | 0
  MCV, Decrease to Low | 1 | 2
  MCV, Change to Normal or No Change | 2 | 2
  MCV, Increase to High | 1 | 0
  Erythrocytes, Decrease to Low | 0 | 0
  Erythrocytes, Change to Normal or No Change | 4 | 4
  Erythrocytes, Increase to High | 0 | 0
  Hematocrit, Decrease to Low | 0 | 0
  Hematocrit, Change to Normal or No Change | 4 | 4
  Hematocrit, Increase to High | 0 | 0
  Monocytes, Decrease to Low | 0 | 0
  Monocytes, Change to Normal or No Change | 2 | 4
  Monocytes, Increase to High | 2 | 0
  Reticulocytes, Decrease to Low | 2 | 1
  Reticulocytes, Change to Normal or No Change | 1 | 3
  Reticulocytes, Increase to High | 1 | 1

12. Primary Outcome: Part 2: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: as for outcome 10
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Anemia, Any Grade Increase | 3 | 3
  Anemia, Increase to Grade 3 | 1 | 1
  Anemia, Increase to Grade 4 | 0 | 0
  Hemoglobin increased, Any Grade Increase | 0 | 0
  Hemoglobin increased, Increase to Grade 3 | 0 | 0
  Hemoglobin increased, Increase to Grade 4 | 0 | 0
  Leukocytosis, Any Grade Increase | 0 | 0
  Leukocytosis, Increase to Grade 3 | 0 | 0
  Leukocytosis, Increase to Grade 4 | 0 | 0
  White blood cell decreased, Any Grade Increase | 2 | 3
  White blood cell decreased, Increase to Grade 3 | 1 | 1
  White blood cell decreased, Increase to Grade 4 | 0 | 1
  Lymphocyte count decreased, Any Grade Increase | 3 | 4
  Lymphocyte count decreased, Increase to Grade 3 | 2 | 1
  Lymphocyte count decreased, Increase to Grade 4 | 0 | 0
  Lymphocyte count increased, Any Grade Increase | 1 | 1
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0
  Neutrophils, Any Grade Increase | 1 | 4
  Neutrophils, Increase to Grade 3 | 0 | 0
  Neutrophils, Increase to Grade 4 | 0 | 2
  Platelets, Any Grade Increase | 3 | 4
  Platelets, Increase to Grade 3 | 1 | 1
  Platelets, Increase to Grade 4 | 2 | 1

13. Primary Outcome: Part 2: Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: Basophils, Eosinophils, MCHC, MCH, MCV, erythrocytes, Hematocrit, monocytes and reticulocytes. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low, changes to normal or no changes, and increases to high from baseline values have been presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Basophils, Decrease to Low | 0 | 0
  Basophils, Change to Normal or No Change | 3 | 1
  Basophils, Increase to High | 0 | 3
  Eosinophils, Decrease to Low | 0 | 0
  Eosinophils, Change to Normal or No Change | 3 | 3
  Eosinophils, Increase to High | 0 | 1
  Hematocrit, Decrease to Low | 1 | 1
  Hematocrit, Change to Normal or No Change | 2 | 3
  Hematocrit, Increase to High | 0 | 0
  MCH, Decrease to Low | 2 | 2
  MCH, Change to Normal or No Change | 1 | 2
  MCH, Increase to High | 1 | 0
  MCHC, Decrease to Low | 0 | 2
  MCHC, Change to Normal or No Change | 3 | 1
  MCHC, Increase to High | 0 | 1
  MCV, Decrease to Low | 1 | 1
  MCV, Change to Normal or No Change | 0 | 2
  MCV, Increase to High | 2 | 1
  Monocytes, Decrease to Low | 0 | 0
  Monocytes, Change to Normal or No Change | 1 | 0
  Monocytes, Increase to High | 2 | 4
  Erythrocytes, Decrease to Low | 0 | 1
  Erythrocytes, Change to Normal or No Change | 3 | 3
  Erythrocytes, Increase to High | 0 | 0
  Reticulocytes, Decrease to Low | 1 | 1
  Reticulocytes, Change to Normal or No Change | 1 | 1
  Reticulocytes, Increase to High | 1 | 2

14. Primary Outcome: Part 1: Number of Participants With Worst-case Change in Post Baseline Values Relative to Baseline Urinalysis Results: Occult Blood and Protein
Description: Urine samples were collected to analyze presence of occult blood and protein in urine by dipstick method. Data for worst-case post baseline urinalysis results is presented. Result for urinalysis parameters were recorded as no change/decreased, Increase to SMALL, Increase to MODERATE, Increase to LARGE, and any increase including increase to +-, 1+, 2+, 3+, unknown indicating proportional concentrations in the urine sample.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population. Only those participants with data available at specified category have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 4 | 2
  Occult Blood, No Change/Decreased | 4 | 2
  Occult Blood, Increase to SMALL: number analyzed (Participants) | 4 | 2
  Occult Blood, Increase to SMALL | 0 | 0
  Occult Blood, Increase to MODERATE: number analyzed (Participants) | 4 | 2
  Occult Blood, Increase to MODERATE | 0 | 0
  Occult Blood, Increase to LARGE: number analyzed (Participants) | 4 | 2
  Occult Blood, Increase to LARGE | 0 | 0
  Protein, No Change/Decreased: number analyzed (Participants) | 4 | 3
  Protein, No Change/Decreased | 2 | 2
  Protein, Increase to +-: number analyzed (Participants) | 4 | 3
  Protein, Increase to +- | 0 | 0
  Protein, Increase to 1+: number analyzed (Participants) | 4 | 3
  Protein, Increase to 1+ | 1 | 1
  Protein, Increase to 2+: number analyzed (Participants) | 4 | 3
  Protein, Increase to 2+ | 1 | 0
  Protein, Increase to 3+: number analyzed (Participants) | 4 | 3
  Protein, Increase to 3+ | 0 | 0
  Protein, Unknown | 0 | 0

15. Primary Outcome: Part 2: Number of Participants With Worst-case Change in Post Baseline Values Relative to Baseline Urinalysis Results: Occult Blood and Protein
Description: as for outcome 14
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified category have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Occult Blood, No Change/Decreased | 3 | 4
  Occult Blood, Increase to SMALL | 0 | 0
  Occult Blood, Increase to MODERATE | 0 | 0
  Occult Blood, Increase to LARGE | 0 | 0
  Protein, No Change/Decreased: number analyzed (Participants) | 3 | 3
  Protein, No Change/Decreased | 1 | 3
  Protein, Increase to +-: number analyzed (Participants) | 3 | 3
  Protein, Increase to +- | 1 | 0
  Protein, Increase to 1+: number analyzed (Participants) | 3 | 3
  Protein, Increase to 1+ | 0 | 0
  Protein, Increase to 2+: number analyzed (Participants) | 3 | 3
  Protein, Increase to 2+ | 0 | 0
  Protein, Increase to 3+: number analyzed (Participants) | 3 | 3
  Protein, Increase to 3+ | 0 | 0
  Protein, Unknown | 1 | 0

16. Primary Outcome: Part 1: Change From Baseline (CFB) in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze urine pH levels. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
pH
  Baseline (Day 1) | 7.13 (0.750) | 5.38 (0.479)
  CFB to 141 Weeks: number analyzed (Participants) | 4 | 3
  CFB to 141 Weeks | -0.75 (0.645) | 0.67 (1.155)

17. Primary Outcome: Part 2: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: as for outcome 16
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
pH
  Baseline (Day 1) | 6.33 (1.041) | 5.25 (0.500)
  CFB to 212 weeks: number analyzed (Participants) | 1 | 2
  CFB to 212 weeks | 0.00 | 1.50 (0.707)

18. Primary Outcome: Part 1: Change From Baseline in Urine Specific Gravity by Dipstick
Description: Urine samples were collected to analyze urine specific gravity. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Ratio
  Baseline (Day 1) | 1.0128 (0.00591) | 1.0190 (0.00408)
  CFB to 141 Weeks: number analyzed (Participants) | 4 | 3
  CFB to 141 Weeks | -0.0010 (0.01010) | -0.0037 (0.00451)

19. Primary Outcome: Part 2: Change From Baseline in Urine Specific Gravity by Dipstick
Description: as for outcome 18
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Ratio
  Baseline (Day 1) | 1.0167 (0.00723) | 1.0218 (0.00608)
  CFB to 212 Weeks: number analyzed (Participants) | 1 | 2
  CFB to 212 Weeks | -0.0070 | -0.0055 (0.00354)

20. Primary Outcome: Part 1: Number of Participants With Worst-case Grade Change Post-baseline in Vital Sign Parameters: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured after resting for at least 5 minutes in a supine or semi-recumbent position. They were graded according to NCI-CTCAE version 4.03. For SBP: Grade (G) 0 (<120 millimeter of mercury [mmHg]), G1 (120-139 mmHg), G2 (140-159 mmHg), G3 (>=160 mmHg). For DBP: G0 (<80 mmHg), G1 (80-89 mmHg), G2 (90-99 mmHg), G3 (>=100 mmHg). Higher grade indicates greater severity. Data for participants with worst-case post baseline with any grade increase and a maximum post-baseline grade increase to G2 and G3 from their baseline grade are presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  SBP, Any Grade Increase | 3 | 2
  SBP, Increase to Grade 2 | 2 | 1
  SBP, Increase to Grade 3 | 1 | 0
  DBP, Any Grade Increase | 2 | 2
  DBP, Increase to Grade 2 | 1 | 0
  DBP, Increase to Grade 3 | 1 | 0

21. Primary Outcome: Part 2: Number of Participants With Worst-case Grade Change Post-baseline in Vital Sign Parameters: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: as for outcome 20
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  SBP, Any Grade Increase | 2 | 2
  SBP, Increase to Grade 2 | 2 | 1
  SBP, Increase to Grade 3 | 0 | 1
  DBP, Any Grade Increase | 2 | 3
  DBP, Increase to Grade 2 | 1 | 2
  DBP, Increase to Grade 3 | 1 | 0

22. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Vital Sign Parameters: Temperature
Description: Temperature was measured after resting for at least 5 minutes. The abnormal ranges for body temperature were (<=35 degrees Celsius or >=38 degrees Celsius). Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Decrease to =<35 | 0 | 0
  Change to Normal or to No Change | 4 | 4
  Increase to >=38 | 0 | 0

23. Primary Outcome: Part 2: Number of Participants With Worst-case Change Post-baseline in Vital Sign Parameters: Temperature
Description: as for outcome 22
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Decrease to <=35 | 0 | 0
  Change to Normal or No Change | 3 | 4
  Increase to >=38 | 0 | 0

24. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Vital Sign Parameters: Heart Rate
Description: Heart rate was measured after resting for at least 5 minutes. The abnormal ranges for heart rate were (low <60 beats per minute [bpm] and high >100 bpm). Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits. Data for participants with worst case change from baseline was presented as Baseline to low, Baseline to Normal or No change and Baseline to High.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Decrease to Low (<60 bpm) | 1 | 0
  Change to Normal or No Change | 3 | 3
  Increase to High (>100 bpm) | 0 | 1

25. Primary Outcome: Part 2: Number of Participants With Worst-case Change Post-baseline in Vital Sign Parameters: Heart Rate
Description: as for outcome 24
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants
  Decrease to Low (<60 bpm) | 1 | 1
  Change to Normal or No Change | 0 | 3
  Increase to High (>100 bpm) | 2 | 0

26. Primary Outcome: Part 1: Number of Participants With Worst-Case Amount of Increase From Baseline Value in Corrected QT Interval Using Fredericia's Formula (QTcF)
Description: 12-lead electrocardiogram (ECG) was obtained using an automated ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QT interval corrected using Fridericia's formula (QTcF) intervals. Grade 0 (<450 millisecond (msec)), Grade 1 (450-480 msec), Grade 2 (481-500 msec), and Grade 3 (≥501 msec). Higher grade indicates greater severity. Data for participants with worst-case post baseline with any grade increase and a post-baseline grade increase to G2 and G3 from their baseline grade are presented. Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  Any Grade Increase | 1 | 0
  Increase to Grade 2 (481 - 500 msec)) | 1 | 0
  Increase to Grade 3 (>= 501 msec)) | 0 | 0

27. Primary Outcome: Part 2: Number of Participants With Worst-Case Amount of Increase From Baseline Value in QTcF
Description: as for outcome 26
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 2 | 2
Participants
  Any Grade Increase | 0 | 0
  Increase to Grade 2 (481 - 500 msec) | 0 | 0
  Increase to Grade 3 (>= 501 msec) | 0 | 0

28. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The number of participants with worst-case post baseline performance status have been presented as 0-5. Where, 0- Fully active; 1- Restricted in strenuous activity but able to carry out light work activities; 2- Capable of self-care but unable to carry out any work activities; 3- Capable of limited self care, confined to bed/chair more than 50% of waking hours; 4- Completely disabled; can't carry on any self care; totally confined to bed/chair and 5- Dead.Baseline was defined as the latest pre-dose assessment within 21 days prior to first dose with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 141 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  0 | 0 | 1
  1 | 3 | 2
  2 | 1 | 0
  3 | 0 | 0
  4-5 | 0 | 0

29. Secondary Outcome: Part 1: Area Under the Concentration-time Curve During the Dosing Interval (AUC (0-tau)) Following Single Dose Administration of Belantamab Mafodotin (Antibody-drug Conjugate (ADC))
Description: Blood samples were collected for pharmacokinetic (PK) analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; End of Infusion (EOI); 1 hour (h), 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic (PK) population included all participants in all treated population from whom at least one PK sample was obtained, analyzed, and was measurable. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/millilitre (h*ug/mL)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Hour*microgram/millilitre (h*ug/mL) | 3694.5965 (26.33) | 3807.9179 (41.80)

30. Secondary Outcome: Part 1: AUC Extrapolated to Infinity (AUC (0-inf)) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
h*ug/mL | 4177.9497 (28.48) | 4243.1678 (48.78)

31. Secondary Outcome: Part 1: AUC From Time Zero to the Time of the Last Quantifiable Concentration (AUC (0 - Tlast)) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
h*ug/mL | 3606.0173 (22.64) | 2392.2534 (128.99)

32. Secondary Outcome: Part 1: Systemic Clearance (CL) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
milliliter per hour (mL/h) | 35.026301 (37.38) | 45.340473 (37.25)

33. Secondary Outcome: Part 1: Apparent Terminal Half-life (t1/2) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Day | 7.373 [6.92 to 8.38] | 7.779 [5.44 to 9.26]

34. Secondary Outcome: Part 1: Terminal Phase Rate Constant (Lambda_z) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (h)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
1/hour (h) | 0.00385688 (8.96) | 0.00394671 (27.64)

35. Secondary Outcome: Part 1: Volume of Distribution at Steady State (Vss) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Liter (L) | 7.475899 (29.10) | 8.216505 (36.05)

36. Secondary Outcome: Part 1: Time of Last Observed Quantifiable Concentration (Tlast) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Day | 21.578 [15.14 to 22.12] | 21.079 [1.00 to 22.03]

37. Secondary Outcome: Part 1: Time to Maximum Plasma Concentration (Tmax) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
hour (h) | 2.600 [1.58 to 3.68] | 1.635 [0.67 to 1.68]

38. Secondary Outcome: Part 1: Concentration at the End of Infusion (C-EOI) Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL
  CYCLE 1 | 30.28 (24.32) | 39.42 (14.15)
  CYCLE 2: number analyzed (Participants) | 3 | 2
  CYCLE 2 | 32.52 (14.13) | 31.44 (58.71)
  CYCLE 3: number analyzed (Participants) | 2 | 1
  CYCLE 3 | 23.25 (20.83) | 32.20
  CYCLE 6: number analyzed (Participants) | 1 | 2
  CYCLE 6 | 23.60 | 29.22 (24.69)
  CYCLE 9: number analyzed (Participants) | 1 | 0
  CYCLE 9 | 24.50 |
  CYCLE 12: number analyzed (Participants) | 0 | 1
  CYCLE 12 |  | 34.50

39. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL
  CYCLE 1 | 36.35 (19.12) | 41.25 (12.80)
  CYCLE 2: number analyzed (Participants) | 3 | 2
  CYCLE 2 | 32.52 (14.13) | 31.44 (58.71)
  CYCLE 3: number analyzed (Participants) | 2 | 1
  CYCLE 3 | 23.25 (20.83) | 32.20
  CYCLE 6: number analyzed (Participants) | 1 | 2
  CYCLE 6 | 23.60 | 29.22 (24.69)
  CYCLE 9: number analyzed (Participants) | 1 | 0
  CYCLE 9 | 24.50 |
  CYCLE 12: number analyzed (Participants) | 0 | 1
  CYCLE 12 |  | 34.50

40. Secondary Outcome: Part 1: Trough Plasma Concentration (Ctrough) Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 5, Cycle 8 and Cycle 11
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 3
ug/mL
  CYCLE 1 | 1.45 (29.42) | 1.39 (109.19)
  CYCLE 2: number analyzed (Participants) | 2 | 1
  CYCLE 2 | 2.41 (75.30) | 1.76
  CYCLE 5: number analyzed (Participants) | 1 | 1
  CYCLE 5 | 3.17 | 2.20
  CYCLE 8: number analyzed (Participants) | 1 | 0
  CYCLE 8 | 3.60 |
  CYCLE 11: number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Part 1: AUC (0-tau) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/millilitre (h*ug/mL)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 3
Hour*microgram/millilitre (h*ug/mL) | 6358.4427 (33.08) | 7143.7202 (45.60)

42. Secondary Outcome: Part 1: AUC (0-inf) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 2
h*ug/mL | 6939.1227 (31.13) | 6789.2291 (11.80)

43. Secondary Outcome: Part 1: AUC (0 - Tlast) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
h*ug/mL | 5839.2501 (32.96) | 4046.1161 (179.35)

44. Secondary Outcome: Part 1: Systemic Clearance (CL) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 2
mL/h | 22.017014 (34.80) | 25.916718 (25.61)

45. Secondary Outcome: Part 1: t1/2 Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 2
Day | 10.046 [6.92 to 10.57] | 9.512 [7.46 to 11.56]

46. Secondary Outcome: Part 1: Lambda_z Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 2
1/h | 0.00319945 (23.42) | 0.00310928 (31.74)

47. Secondary Outcome: Part 1: Vss Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 3 | 2
Liter (L) | 6.390107 (18.84) | 6.718238 (59.09)

48. Secondary Outcome: Part 1: Tlast Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: day
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
day | 18.627 [14.08 to 22.12] | 21.079 [1.00 to 22.03]

49. Secondary Outcome: Part 1: Tmax Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
hour (h) | 2.695 [1.62 to 8.53] | 1.675 [0.63 to 3.65]

50. Secondary Outcome: Part 1: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL
  CYCLE 1 | 32.68 (27.15) | 45.65 (8.62)
  CYCLE 2: number analyzed (Participants) | 3 | 2
  CYCLE 2 | 38.17 (17.01) | 40.97 (14.90)
  CYCLE 3: number analyzed (Participants) | 2 | 1
  CYCLE 3 | 35.56 (18.19) | 46.10
  CYCLE 6: number analyzed (Participants) | 1 | 2
  CYCLE 6 | 32.00 | 39.14 (19.27)
  CYCLE 9: number analyzed (Participants) | 1 | 0
  CYCLE 9 | 40.90 |
  CYCLE 12: number analyzed (Participants) | 0 | 1
  CYCLE 12 |  | 36.60

51. Secondary Outcome: Part 1: Cmax Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL
  CYCLE 1 | 39.51 (17.00) | 48.89 (14.07)
  CYCLE 2: number analyzed (Participants) | 3 | 2
  CYCLE 2 | 38.17 (17.01) | 40.97 (14.90)
  CYCLE 3: number analyzed (Participants) | 2 | 1
  CYCLE 3 | 35.56 (18.19) | 46.10
  CYCLE 6: number analyzed (Participants) | 1 | 2
  CYCLE 6 | 32.00 | 39.14 (19.27)
  CYCLE 9: number analyzed (Participants) | 1 | 0
  CYCLE 9 | 40.90 |
  CYCLE 12: number analyzed (Participants) | 0 | 1
  CYCLE 12 |  | 36.60

52. Secondary Outcome: Part 1: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 5, Cycle 8 and Cycle 11
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 2 | 3
ug/mL
  CYCLE 1 | 4.47 (22.16) | 5.19 (104.06)
  CYCLE 2: number analyzed (Participants) | 2 | 1
  CYCLE 2 | 6.34 (87.45) | 6.07
  CYCLE 5: number analyzed (Participants) | 1 | 2
  CYCLE 5 | 11.40 | 4.04 (152.78)
  CYCLE 8: number analyzed (Participants) | 1 | 0
  CYCLE 8 | 18.10 |
  CYCLE 11: number analyzed (Participants) | 0 | 1
  CYCLE 11 |  | 1.37

53. Secondary Outcome: Part 1: AUC (0 - Tlast) Following Single Dose Administration of Belantamab Mafodotin Cysteine Maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
h*ug/mL | 73.3412 (44.73) | 141.9031 (77.03)

54. Secondary Outcome: Part 1: Cmax Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL | 748.94 (30.49) | 2797.27 (326.50)

55. Secondary Outcome: Part 1: Tlast Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: day
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
day | 6.940 [6.84 to 14.89] | 6.930 [1.00 to 7.02]

56. Secondary Outcome: Part 1: Tmax Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose; EOI; 1 h, 3 h, 8 h and 24 h post-EOI, Day 8, Day 15 in Cycle 1; Pre-Dose on Cycle 2 Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
hour (h) | 16.380 [8.55 to 24.58] | 16.240 [8.45 to 24.10]

57. Secondary Outcome: Part 1: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL
  CYCLE 1 | 304.99 (61.67) | 330.71 (23.09)
  CYCLE 2: number analyzed (Participants) | 3 | 2
  CYCLE 2 | 195.09 (12.59) | 221.76 (31.09)
  CYCLE 3: number analyzed (Participants) | 2 | 1
  CYCLE 3 | 270.80 (57.38) | 222.00
  CYCLE 6: number analyzed (Participants) | 1 | 2
  CYCLE 6 | 288.80 | 205.70 (13.62)
  CYCLE 9: number analyzed (Participants) | 1 | 0
  CYCLE 9 | 222.80 |
  CYCLE 12: number analyzed (Participants) | 0 | 1
  CYCLE 12 |  | 234.90

58. Secondary Outcome: Part 1: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 5, Cycle 8 and Cycle 11
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
ug/mL | NA (NA) — Due to shorter half-life of cys-mcMMAF, the concentration values were below the Lower Limit of Quantification (LLOQ). Hence, Ctrough values were not determined. | NA (NA) — Due to shorter half-life of cys-mcMMAF, the concentration values were below the Lower Limit of Quantification (LLOQ). Hence, Ctrough values were not determined.

59. Secondary Outcome: Part 1: Observed Accumulation Ratio of C-EOI (R(C-EOI)) Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. Accumulation ratio for C-EOI was calculated as C-EOI at the visit divided by C-EOI at Cycle 1.
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed. Values were not calculated for some cycles since there were no sufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 2 | 1
Ratio | 0.783 (16) | 0.925

60. Secondary Outcome: Part 1: Observed Accumulation Ratio of Ctrough (R(Ctrough)) Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. Accumulation ratio for Ctrough was calculated as Ctrough at the visit divided by pre-dose at Cycle 2 Day 1.
Time Frame: Cycle 1, Cycle 2, Cycle 5, Cycle 8 and Cycle 11
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 2 | 1
Ratio | 1.561 (30) | 1.909

61. Secondary Outcome: Part 1: Observed Accumulation Ratio of C-EOI (R(C-EOI)) Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: as for outcome 59
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 2 | 1
Ratio | 1.139 (26) | 1.075

62. Secondary Outcome: Part 1: Observed Accumulation Ratio of Ctrough (R(Ctrough)) Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: as for outcome 60
Time Frame: Cycle 1, Cycle 2, Cycle 5, Cycle 8 and Cycle 11
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 1 | 1
Ratio | 2.069 | 1.775

63. Secondary Outcome: Part 1: Observed Accumulation Ratio of C-EOI (R(C-EOI)) Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: as for outcome 59
Time Frame: Cycle 1, Cycle 2, Cycle 3, Cycle 6, Cycle 9 and Cycle 12
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 2 | 1
Ratio | 0.603 (117) | 0.869

64. Secondary Outcome: Part 2: AUC (0-tau) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, EOI, 2h and 24h post- Start of Infusion (SOI), Day 4, Day 8-15 in Cycle 1; Pre-Dose on Cycle 2 Day 1 (If Cycle 2 belantamab mafodotin dose was delayed, 1 PK sample was taken at 21 days post-SOI in Arm A or 28 days post-SOI in Arm B)
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h*ug/mL | 5077.3323 (13.10) | 5489.6508 (25.39)

65. Secondary Outcome: Part 2: AUC (0-inf) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 2 | 3
h*ug/mL | 6201.7657 (18.62) | 6178.4350 (30.75)

66. Secondary Outcome: Part 2: AUC (0 - Tlast) Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h*ug/mL | 5160.2733 (10.83) | 5166.5353 (31.90)

67. Secondary Outcome: Part 2: CL Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 2 | 3
mL/h | 24.684617 (4.44) | 20.900323 (7.20)

68. Secondary Outcome: Part 2: Cmax Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
ug/mL | 47.62 (25.07) | 61.70 (26.51)

69. Secondary Outcome: Part 2: Lambda_z Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
1/h | 0.00302685 (15.54) | 0.00470710 (59.70)

70. Secondary Outcome: Part 2: Vss Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 2 | 3
Liter (L) | 6.801065 (4.67) | 4.537404 (22.01)

71. Secondary Outcome: Part 2: t1/2 Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Day | 8.825 [8.63 to 11.40] | 6.195 [3.09 to 11.95]

72. Secondary Outcome: Part 2: Tlast Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Day | 21.080 [20.99 to 24.14] | 27.958 [6.93 to 27.98]

73. Secondary Outcome: Part 2: Tmax Following Single Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
hour (h) | 0.780 [0.72 to 1.85] | 1.865 [0.82 to 2.20]

74. Secondary Outcome: Part 2 Arm A: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 4, Cycle 6, Cycle 9, Cycle 10, Cycle 11 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 3
ug/mL
  CYCLE 1 | 46.34 (27.07)
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 34.80
  CYCLE 6: number analyzed (Participants) | 1
  CYCLE 6 | 47.20
  CYCLE 9: number analyzed (Participants) | 1
  CYCLE 9 | 35.90
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 48.20
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 25.60
  CYCLE 12: number analyzed (Participants) | 1
  CYCLE 12 | 37.60

75. Secondary Outcome: Part 2 Arm A: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 3, Cycle 5, Cycle 8, Cycle 9, Cycle 10 and Cycle 11
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed. Ctrough values were not determined for cycles where the concentration values were below the Lower Limit of Quantification (LLOQ).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 1
ug/mL
  CYCLE 3 | 0.56
  CYCLE 5: number analyzed (Participants) | 0
  CYCLE 8: number analyzed (Participants) | 0
  CYCLE 9: number analyzed (Participants) | 0
  CYCLE 10: number analyzed (Participants) | 0
  CYCLE 11: number analyzed (Participants) | 0

76. Secondary Outcome: Part 2 Arm B: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 4, Cycle 10, Cycle 11 and Cycle 24
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 4
ug/mL
  CYCLE 1 | 52.96 (21.31)
  CYCLE 2: number analyzed (Participants) | 1
  CYCLE 2 | 34.30
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 53.90
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 52.10
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 45.70
  CYCLE 24: number analyzed (Participants) | 1
  CYCLE 24 | 32.00

77. Secondary Outcome: Part 2 Arm B: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (ADC)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 3, Cycle 9, Cycle 10 and Cycle 23
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 1
ug/mL
  CYCLE 1 | 1.05
  CYCLE 3: number analyzed (Participants) | 0
  CYCLE 9: number analyzed (Participants) | 0
  CYCLE 10: number analyzed (Participants) | 0
  CYCLE 23: number analyzed (Participants) | 0

78. Secondary Outcome: Part 2: AUC (0-tau) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h*ug/mL | 9213.7145 (6.50) | 9590.8606 (23.71)

79. Secondary Outcome: Part 2: AUC (0-inf) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed. AUC(0-inf) were not calculated for some participants since there were no sufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 0 | 2
h*ug/mL |  | 9921.8634 (11.55)

80. Secondary Outcome: Part 2: AUC (0 - Tlast) Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h*ug/mL | 9471.9799 (1.97) | 8495.7663 (36.72)

81. Secondary Outcome: Part 2: Cmax Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
ug/mL | 43.51 (15.05) | 52.33 (22.64)

82. Secondary Outcome: Part 2: Lambda_z Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
1/h | 0.00159877 (22.83) | 0.00305831 (45.34)

83. Secondary Outcome: Part 2: Vss Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed. Vss was not calculated for some participants as sufficient data was not available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 0 | 2
Liter (L) |  | 4.367635 (9.29)

84. Secondary Outcome: Part 2: t1/2 Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Day | 16.172 [15.57 to 23.41] | 10.392 [5.18 to 14.30]

85. Secondary Outcome: Part 2: Tlast Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Day | 21.080 [20.99 to 24.14] | 27.958 [6.93 to 27.98]

86. Secondary Outcome: Part 2: Tmax Following Single Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
hour (h) | 1.850 [1.75 to 2.20] | 1.900 [1.75 to 2.20]

87. Secondary Outcome: Part 2: Arm A: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 4, Cycle 6, Cycle 9, Cycle 10, Cycle 11 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 3
ug/mL
  CYCLE 1 | 40.80 (10.98)
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 40.80
  CYCLE 6: number analyzed (Participants) | 1
  CYCLE 6 | 38.20
  CYCLE 9: number analyzed (Participants) | 1
  CYCLE 9 | 43.60
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 55.70
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 30.40
  CYCLE 12: number analyzed (Participants) | 1
  CYCLE 12 | 35.20

88. Secondary Outcome: Part 2: Arm A: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 3, Cycle 5, Cycle 8, Cycle 9, Cycle 10 and Cycle 11
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 1
ug/mL
  CYCLE 3 | 2.11
  CYCLE 5 | 0.84
  CYCLE 8 | 1.77
  CYCLE 9: number analyzed (Participants) | 0
  CYCLE 10 | 1.41
  CYCLE 11 | 0.74

89. Secondary Outcome: Part 2: Arm B: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 4, Cycle 10, Cycle 11 and Cycle 24
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3
ug/mL
  CYCLE 1 | 55.85 (12.63)
  CYCLE 2: number analyzed (Participants) | 1
  CYCLE 2 | 42.40
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 46.30
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 54.00
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 71.40
  CYCLE 24: number analyzed (Participants) | 1
  CYCLE 24 | 34.30

90. Secondary Outcome: Part 2: Arm B: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Total Antibody)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 3, Cycle 9, Cycle 10 and Cycle 23
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 1
ug/mL
  CYCLE 1 | 4.14
  CYCLE 3: number analyzed (Participants) | 0
  CYCLE 9 | 3.09
  CYCLE 10: number analyzed (Participants) | 0
  CYCLE 23 | 0.82

91. Secondary Outcome: Part 2: AUC (0 - Tlast) Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nanogram (ng)/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h*nanogram (ng)/mL | 80.0859 (22.53) | 82.6253 (42.28)

92. Secondary Outcome: Part 2: Cmax Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram (pg)/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
picogram (pg)/mL | 857.63 (32.99) | 905.42 (28.37)

93. Secondary Outcome: Part 2: Tlast Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Day
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Day | 6.942 [6.81 to 7.01] | 6.865 [3.90 to 7.79]

94. Secondary Outcome: Part 2: Tmax Following Single Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 64
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: h
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
h | 22.370 [22.05 to 23.07] | 22.950 [22.03 to 24.15]

95. Secondary Outcome: Part 2 Arm A: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 4, Cycle 6, Cycle 9, Cycle 10, Cycle 11 and Cycle 12
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 3
pg/mL
  CYCLE 1 | 319.85 (29.78)
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 399.10
  CYCLE 6: number analyzed (Participants) | 1
  CYCLE 6 | 207.50
  CYCLE 9: number analyzed (Participants) | 1
  CYCLE 9 | 88.60
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 179.00
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 232.00
  CYCLE 12: number analyzed (Participants) | 1
  CYCLE 12 | 336.00

96. Secondary Outcome: Part 2: Arm A: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 3, Cycle 5, Cycle 8, Cycle 9, Cycle 10 and Cycle 11
Population: Pharmacokinetic population. Due to shorter half-life of cys-mcMMAF, the concentration values were below the Lower Limit of Quantification (LLOQ). Hence, Ctrough values were not determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex)
Number analyzed (Participants) | 3

97. Secondary Outcome: Part 2: Arm B: C-EOI Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 2, Cycle 4, Cycle 10, Cycle 11 and Cycle 24
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 4
pg/mL
  CYCLE 1 | 390.28 (46.28)
  CYCLE 2: number analyzed (Participants) | 1
  CYCLE 2 | 428.60
  CYCLE 4: number analyzed (Participants) | 1
  CYCLE 4 | 499.80
  CYCLE 10: number analyzed (Participants) | 1
  CYCLE 10 | 198.00
  CYCLE 11: number analyzed (Participants) | 1
  CYCLE 11 | 269.00
  CYCLE 24: number analyzed (Participants) | 1
  CYCLE 24 | 346.00

98. Secondary Outcome: Part 2: Arm B: Ctrough Following Repeat Dose Administration of Belantamab Mafodotin (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Cycle 1, Cycle 3, Cycle 9, Cycle 10 and Cycle 23
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 4
pg/mL | NA (NA) — Due to shorter half-life of cys-mcMMAF, the concentration values were below the Lower Limit of Quantification (LLOQ). Hence, Ctrough values were not determined.

99. Secondary Outcome: Part 1: Number of Participants With Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples were collected and tested for the presence of antibodies against belantamab mafodotin.
Time Frame: Up to approximately 141 weeks
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

100. Secondary Outcome: Part 2: Number of Participants With Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples were collected and tested for the presence of antibodies against belantamab mafodotin.
Time Frame: Up to approximately 212 weeks
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

101. Secondary Outcome: Part 1: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to approximately 141 weeks
Population: All Treated Population. There were no participants with positive ADA results. Hence the titer (concentration) of ADA was not collected.
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 0 | 0

102. Secondary Outcome: Part 2: Titers of ADAs Against Belantamab Mafodotin
Description: as for outcome 101
Time Frame: Up to approximately 212 weeks
Population: as for outcome 101
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 0 | 0

103. Secondary Outcome: Part 1 - Percentage of Participants With Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed partial response (PR) or better (i.e. PR, very good partial response [VGPR], complete response [CR], and stringent complete response [sCR]) of best response, according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR= CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-component plus urine M-component <100 mg/24 hour (h); PR = >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 h.
Time Frame: Up to approximately 141 weeks
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Percentage of Participants | 50 [6.8 to 93.2] | 25 [0.6 to 80.6]

104. Secondary Outcome: Part 2 - Percentage of Participants With ORR
Description: ORR is defined as the percentage of participants with a confirmed PR or better (i.e. PR, VGPR, CR, and sCR) of best response, according to the IMWG Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR= CR as above PLUS normal serum FLC assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = >=50% reduction of serum M-protein and reduction in 24-h urinary M-protein by >=90% or to <200 mg/24 h.
Time Frame: Up to approximately 212 weeks
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Percentage of Participants | 100 [29.2 to 100.0] | 50 [6.8 to 93.2]

105. Secondary Outcome: Part 1: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of participants with a confirmed Minimal response (MR) or better (i.e. MR, PR, VGPR, CR, and sCR) of best response, according to the IMWG Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR= CR as above PLUS normal serum FLC assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = >=50% reduction of serum M-protein and reduction in 24-h urinary M-protein by >=90% or to <200 mg/24 h; MR= >=25% but <=49% reduction of serum M-protein and reduction in 24-h urine M-protein by 50-89%. In addition to the above listed criteria, if present at baseline, >=50% reduction in the size (SPD) 4 of soft tissue plasmacytomas is also required.
Time Frame: Up to approximately 141 weeks
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg
Number analyzed (Participants) | 4 | 4
Percentage of Participants | 50 [6.8 to 93.2] | 75 [19.4 to 99.4]

106. Secondary Outcome: Part 2: Clinical Benefit Rate (CBR)
Description: as for outcome 105
Time Frame: Up to approximately 212 weeks
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Percentage of Participants | 100 [29.2 to 100.0] | 50 [6.8 to 93.2]

107. Primary Outcome: Part 2: Number of Participants With Clinically Significant Abnormalities in ECOG Performance Status
Description: Any change in ECOG Performance status that was clinically significant in the medical and scientific judgment of the investigator and not related to an underlying disease was reported.
Time Frame: Baseline (Day 1) and up to approximately 212 weeks
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex)
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 212 weeks for main study and up to approximately 74 weeks for PACT phase.
Description: Safety population included all participants who received at least 1 dose of study treatment.
  MedDRA version 24.1 was used for Part 1 (P1) and 26.0 for Part 2 (P2).
Arm/Group | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex)
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 0/3 | 0/4 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/4 | 0/3 | 1/4 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/3 | 4/4 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) (N=4) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg (N=4) | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) (N=3) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) (N=4) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) (N=2) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex) (N=2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intratumoural haematoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Part 1: Belantamab Mafodotin 2.5 Milligram/ Kilogram (mg/kg) (N=4) | Main Study - Part 1: Belantamab Mafodotin 3.4 mg/kg (N=4) | Main Study - Part 2: ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) (N=3) | Main Study - Part2: ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dexamethasone (Pom/Dex) (N=4) | PACT Phase - ArmA-Belantamab Mafodotin 2.5 mg/kg + Bortezomib and Dexamethasone (Bor/Dex) (N=2) | PACT Phase - ArmB- Belantamab Mafodotin 2.5 mg/kg + Pomalidomide and Dex (Pom/Dex) (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral mucosa erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea nigra (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (19) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (6) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03828292/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03828292/SAP_001.pdf